CLINICAL TRIAL: NCT02698137
Title: Quality Assessment in ERCP: Risk Factors for Procedure-related Complications in Patients Undergoing ERCP in the Setting of an Endoscopy Training Program
Brief Title: Quality Assessment in Endoscopic Retrograde Cholangiopancreatography(ERCP)
Acronym: QUASIE2
Status: Completed | Type: Observational
Sponsor: Clinical Hospital Colentina (Other)
Responsible Party: Principal Investigator, dr. Theodor Alexandru Voiosu, MD, PhD, Clinical Hospital Colentina
Other Study IDs: QUASIE2
Record Dates: First submitted 2016-02-24; First posted 2016-03-03 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde; Common Bile Duct Lithiasis; Biliary Strictures; Bile Duct and Pancreatic Tumors
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will prospectively collect patient and procedure-related data in an observational study in order to detect patient and procedure-related risk factors for poor outcome (i.e. technical failure of the procedure; procedure-related complications).

Data will be prospectively reported using standard report forms and patients will be followed up to 30 days to detect late-onset complications.

DETAILED DESCRIPTION:
This is an investigator-driven, prospective multicenter trial which analyzes the impact of trainee participation on procedure-related outcome (technical success and procedure-related complications).

All ERCPs in the participating centers will be documented using a standard report form which will require the attending endoscopist to provide data relating to the patient (age, gender, diagnosis, bilirubin levels) and the procedure (including but not limited to the indication, technical aspects including cannulation technique, time to cannulation, degree of trainee involvement - where appropriate, procedure-related adverse events and their outcome).

Because teaching ERCP is not yet a standardized procedure, we aim to assemble a large database, stemming from the experience of several teaching centers in order to identify the main patient and operator-related factors which might influence the outcome of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing ERCP with attempted cannulation of either the major or minor papilla

Exclusion Criteria:

* refusal to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all consecutive patients undergoing ERCP in an endoscopy training program setting
Sampling Method: Non-Probability Sample
Enrollment: 1843 (Actual)
Dates: Start 2016-03; Primary Completion 2019-01 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
procedure-related adverse events | 30 days
  the percentage of patients experiencing procedure-related adverse events (i.e post-ERCP pancreatitis; postERCP cholangitis; perforation; postERCP bleeding or death) occuring within 30 days of the procedure

SECONDARY OUTCOMES:
technical failure of the procedure | 30 days
  percentage of procedures where the operator was unable to achieve the desired therapeutic goal (i.e selective cannulation, stone removal, stenting)

CONTACTS AND LOCATIONS:
Overall Officials: Theodor Voiosu, MD, PhD, Principal Investigator — Clinical Hospital Colentina
Locations (3):
- GI Endoscopy Unit, Department of Gastroenterology and Hepatology, University Hospital Zagreb, Zagreb, Croatia
- Endoscopia Digestiva Chirurgica, Policlinico Gemelli, Roma, Italy
- Gastroenterology Department, Colentina Hospital, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Voiosu TA, Bengus A, Haidar A, Rimbas M, Zlate A, Balanescu P, Voiosu A, Voiosu R, Mateescu B. Antibiotic Prophylaxis Prior to Elective ERCP Does Not Alter Cholangitis Rates or Shorten Hospital Stay: Results of an Observational Prospective Study of 138 Consecutive ERCPS. Maedica (Bucur). 2014 Dec;9(4):328-32. PMID 25705300